CLINICAL TRIAL: NCT01354938
Title: Outcome Study to Evaluate the Role of Klaricid XL (Clarithromycin Modified Release) in the Treatment of Acute Exacerbation of Chronic Bronchitis (AECB) and Its Impact on Quality of Life Measured by St. George's Respiratory Questionnaire (SGRQ)
Brief Title: Outcome Study to Evaluate Klaricid XL® (Clarithromycin Modified Release) in Patients With Acute Exacerbation of Chronic Bronchitis
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: P12-822
Record Dates: First submitted 2011-05-16; First posted 2011-05-17 (Estimated); Results first posted 2013-01-30 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Bronchitis
Keywords: Bronchitis
MeSH Terms: conditions — Bronchitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute Exacerbation of Chronic Bronchitis (AECB): Participants with a diagnosis of chronic bronchitis and signs and symptoms of an acute exacerbation who were prescribed Klaricid XL (500 mg of modified release clarithromycin) at a dose of one tablet once a day or two tablets once a day based on physician's decision of severity of symptoms per routine clinical care.
  Interventions: Drug: Clarithromycin modified release 500 mg

INTERVENTIONS:
Drug: Clarithromycin modified release 500 mg — Clarithromycin modified release 500 mg was prescribed. The dosage given was either 1 tablet or 2 tablets once a day, depending on the severity of the treatment.

SUMMARY:
The objective of this study was to evaluate the role of Klaricid XL (clarithromycin modified release) in the treatment of acute exacerbation of chronic bronchitis (AECB) and its impact on improving the quality of life.

DETAILED DESCRIPTION:
Participants in this observational study had a diagnosis of chronic bronchitis and signs and symptoms of an acute exacerbation, clinically diagnosed by the sudden worsening of symptoms characterized by extreme breathlessness and increased chest tightness, wheezing, cough, or sputum changes. A sequential non-systematic sample of patients with AECB from May 2011 until January 04, 2012 is included in this observational study.

The observation period for each individual patient started with the diagnosis of the acute exacerbation of chronic bronchitis and prescription of antimicrobial medication per routine clinical care. This observational period continued during the treatment period and ended on at least one follow-up visit at the end of the treatment. Duration of treatment was based on physician's judgment of severity of the patient's condition. The usual treatment period ranges from 5 to 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute exacerbation of chronic bronchitis who required antimicrobial therapy and treated with Klaricid XL (clarithromycin modified release)
* Male and female patients age 35 years and older

Exclusion Criteria:

* Patients with clinical signs and symptoms suggesting pneumonia
* Patients with asthma
* Patients with any concomitant illness that may confound the interpretation of the effect of study medication (e.g., pulmonary malignancy, congestive heart failure, bronchiectasis, pneumothorax)
* Immunocompromised patients; however, patients receiving systemic steroids at baseline for the treatment of chronic obstructive pulmonary disease can be enrolled
* Pregnant females
* Nursing mothers
* Patients who are allergic to clarithromycin

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2011-05; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raeef Ahmed, MD, Study Director — Abbott
Locations (28):
- Pakistan (28):
  - Site Ref # / Investigator 54037, Peshawar, Khyber Pakhtunkhwa
  - Site Ref # / Investigator 54044, Multan, Punjab Province
  - Site Ref # / Investigator 54026, Faisalabad
  - Site Ref # / Investigator 54028, Faisalabad
  - Site Ref # / Investigator 54029, Faisalabad
  - Site Ref # / Investigator 54015, Hyderābād
  - Site Ref # / Investigator 54016, Hyderābād
  - Site Ref # / Investigator 54017, Hyderābād
  - Site Ref # / Investigator 54018, Hyderābād
  - Site Ref # / Investigator 54035, Islamabad
  - Site Ref # / Investigator 54002, Karachi
  - Site Ref # / Investigator 54003, Karachi
  - Site Ref # / Investigator 54004, Karachi
  - Site Ref # / Investigator 54005, Karachi
  - Site Ref # / Investigator 54006, Karachi
  - Site Ref # / Investigator 54007, Karachi
  - Site Ref # / Investigator 54009, Karachi
  - Site Ref # / Investigator 54010, Karachi
  - Site Ref # / Investigator 54013, Karachi
  - Site Ref # / Investigator 54019, Lahore
  - Site Ref # / Investigator 54020, Lahore
  - Site Ref # / Investigator 54022, Lahore
  - Site Ref # / Investigator 54023, Lahore
  - Site Ref # / Investigator 54040, Multan
  - Site Ref # / Investigator 54043, Multan
  - Site Ref # / Investigator 55270, Multan
  - Site Ref # / Investigator 55273, Peshawar
  - Site Ref # / Investigator 54033, Rawalpindi

RESULTS

PARTICIPANT FLOW:
Groups:
- Acute Exacerbation of Chronic Bronchitis (AECB): Participants with a diagnosis of chronic bronchitis and signs and symptoms of an acute exacerbation who were prescribed Klaricid XL (500 mg of modified release clarithromycin) at a dose of one tablet once a day or two tablets once a day, based on physician's decision of severity of symptoms, per routine clinical care.
Period: Overall Study
Arm/Group | Acute Exacerbation of Chronic Bronchitis (AECB)
Started | 220
Completed | 219
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Acute Exacerbation of Chronic Bronchitis (AECB)
Number analyzed (Participants) | 220
Age Continuous [Mean (Standard Deviation); unit: years] | 56.35 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 193
Region of Enrollment [Number; unit: participants]
  Pakistan | 220

OUTCOME MEASURES:

1. Primary Outcome: St. George's Respiratory Questionnaire (SGRQ) Scores at Baseline and End of Treatment
Description: The SGRQ is a 50-item questionnaire with 76 weighted responses. It provides a Total score and three component scores: Symptoms (distress caused by respiratory symptoms), Activity (physical activities that cause or are limited by breathlessness), and Impacts (social and psychological effects of the disease). The Total score and each of the SGRQ subscores are scored from 0 to 100 where 0 indicates best and 100 indicates worst health. An increase in score indicates worsening health. A change in the Total score of 4 units is consistent with a clinically significant change in the participant.
Time Frame: Baseline, End of Treatment (maximum treatment duration of 10 days)
Population: Participants with evaluable data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acute Exacerbation of Chronic Bronchitis (AECB)
Number analyzed (Participants) | 219
units on a scale
  Symptoms Score at Baseline | 69.6 (20.0)
  Activity Score at Baseline | 67.4 (20.8)
  Impacts Score at Baseline | 61.0 (22.6)
  Total Score at Baseline | 64.5 (19.2)
  Symptoms Score at End of Treatment | 43.7 (23.2)
  Activity Score at End of Treatment | 51.8 (21.2)
  Impacts Score at End of Treatment | 37.8 (21.0)
  Total Score at End of Treatment | 43.2 (18.9)

2. Secondary Outcome: Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE)
Description: AE=any untoward medical occurrence in a patient, which does not necessarily have a causal relationship with their treatment. SAE=an event meeting any of the following criteria: results in death, hospitalization, prolongation of hospitalization, is life-threatening, congenital anomaly, persistent or significant disability/incapacity, important medical event requiring medical or surgical intervention, spontaneous or elective abortion. AEs and SAEs were collected during the course of the study. See the Reported Adverse Event section for details.
Time Frame: From start of treatment (maximum treatment duration was 10 days) through last follow up visit (3 to 4 weeks after end of treatment)
Population: All enrolled participants
Measure: Number; unit: participants
Arm/Group | Acute Exacerbation of Chronic Bronchitis (AECB)
Number analyzed (Participants) | 220
participants
  Any AE | 12
  Any SAE | 1

3. Primary Outcome: Number of Participants With a Minimal Clinically Important Difference (MCID) in SGRQ Total Score at End of Treatment
Description: The SGRQ is a 50-item questionnaire with 76 weighted responses. It provides a Total score and three component scores: Symptoms (distress caused by respiratory symptoms), Activity (physical activities that cause or are limited by breathlessness), and Impacts (social and psychological effects of the disease). The Total score and each of the SGRQ subscores are scored from 0 to 100 where 0 indicates best and 100 indicates worst health. An increase in score indicates worsening health. The change from Baseline of 4 or more units lower, consistent with a clinically significant change in the participant, was considered in this study to be the 'minimal clinically important difference' (MCID).
Time Frame: Baseline, End of Treatment (maximum treatment duration of 10 days)
Population: Participants with evaluable data
Measure: Number; unit: participants
Arm/Group | Acute Exacerbation of Chronic Bronchitis (AECB)
Number analyzed (Participants) | 219
participants | 176

ADVERSE EVENTS:
Time Frame: From start of treatment (maximum treatment duration was 10 days) through last follow up visit (3 to 4 weeks after end of treatment)
Arm/Group | Acute Exacerbation of Chronic Bronchitis (AECB)
Serious Adverse Events (participants affected / at risk) | 1/220
Other Adverse Events (participants affected / at risk) | 11/220
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Acute Exacerbation of Chronic Bronchitis (AECB) (N=220)
Stevens-Johnson Syndrome (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Acute Exacerbation of Chronic Bronchitis (AECB) (N=220)
Vertigo (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Pruritis generalized (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Dysgeusia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Decreased appetite (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Hypoglycaemia (Endocrine disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.